CLINICAL TRIAL: NCT05835518
Title: An Observational, Prospective Study to Assess the Efficacy and Safety of Adalloce in Patients With Rheumatoid Arthritis and Ankylosing Spondylitis
Brief Title: An Observational, Prospective Study to Assess the Efficacy and Safety of Adalloce in Patients With RA and AS
Status: Recruiting | Type: Observational
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: YMC049
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis
Keywords: The Efficacy and Safety of Adalloce
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This Study is to Assess the Efficacy and Safety of Adalloce in Patients With Rheumatoid Arthritis and Ankylosing Spondylitis, An Observational, Prospective Study

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of over 19 and under 75 at the time of consent
2. Patients diagnosed with RA or AS at least 3 months prior to the study registration
3. Patients who are scheduled to be prescribed Adalloce according to the doctor's opinions
4. Patients who have never received Adalloce
5. Patients who voluntarily gave their written consent after being sufficiently explained about the purpose and contents of this study

Exclusion Criteria:

1. Patients with hypersensitivity to this drug or its components
2. Patients with active tuberculosis or other severe infection such as sepsis or opportunistic infection
3. Patients with moderate to severe heart failure (NYHA class III/IV)
4. Patients who are judged to be inappropriate for Adalloce administration according to the approved conditions
5. Patients who are not suitable for participation in this study according to the judgment of the investigator
6. Patients participating in other drug clinical trials (Adalloce PMS participants cannot participate in this study)

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those diagnosed with RA or AS
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Changes in quality of life (EQ-5D-5L) scores at 52 weeks from baseline in patients with RA and AS | 52weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeongyoon Choi, PI, Principal Investigator — Daegu Catholic University Medical Center
Locations (1):
- Daegu Catholic University Medical Center, Daegu, South Korea